CLINICAL TRIAL: NCT03669484
Title: International Multicenter Single Blind Randomized Clinical Study to Compare Efficacy and Safety of Remimazolam and Propofol in Patients Undergoing Elective Surgical Procedures Under General Anesthesia
Brief Title: Comparative Clinical Study of Efficacy and Safety of Remimazolam and Propofol in Patients Undergoing Elective Surgery Under General Anaesthesia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: R-Pharm (Industry)
Collaborators: Synergy Research Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CN01082020
Record Dates: First submitted 2018-09-07; First posted 2018-09-13 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: General Anaesthesia
Keywords: anaesthesia; surgery
MeSH Terms: interventions — remimazolam; Propofol; Fentanyl; Rocuronium

STUDY DESIGN:
Who Masked: Participant
Masking Description: Simple blinding stipulates hiding the treatment group for a patient. In addition, the research team had a blinded anesthesiologist who did not know about a patient's therapy group throughout the trial. This anesthesiologist assessed a patient's condition by scales (modified Aldrete score, memory assessment, postoperative delirium diagnosis). Anesthesia depth assessment by bispectral index (BIS), administration and, if necessary, correction of the trial drug/reference drug dosage were carried out by another anesthesiologist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remimazolam (Experimental): The induction of anesthesia: intravenous infusion of 6 mg/kg/h until registration of loss of consciousness.
  Maintenance of anesthesia: Remimazolam intravenous infusion initiated at a dose of 1 mg/kg/h; the dose level was adjusted accordingly based on a systemic patient monitoring until the end of operation to 2 mg/kg/h maximum; In case of loss of consciousness was not registered in 2.5 minutes of continuous intravenous infusion: drug administration was terminated. If loss of consciousness was not registered during 30 seconds, other sedative drugs were used for induction and maintenance of anesthesia.
  In case of signs of awakening (fluctuation of blood pressure/heart rate, lacrimation, sweating, etc.) were observed: intravenous bolus infusion (maximum level of 12 mg/kg/h for 1 minute). If signs of awakening remained remimazolam administration was discontinued and other sedatives were used.
  Interventions: Drug: Remimazolam; Drug: Fentanyl; Drug: Rocuronium bromide
- Propofol (Active Comparator): The induction of anesthesia: intravenous infusion of 1.5-2.5 mg/kg for about 1 minute.
  Maintenance of anesthesia: intravenous infusion for a total dose of 4-12 mg/kg/h; the dose level was adjusted accordingly based on a systemic patient monitoring until the end of operation.
  In case of loss of consciousness was not registered other sedative drugs were used for induction and maintenance of anesthesia.
  In case of signs of awakening (fluctuation of blood pressure/heart rate, lacrimation, sweating, etc.) were observed and propofol dose adjustment had not resulted in the desired effect and signs of awakening were saved: the use of propofol was discontinued and other sedatives were used.
  Interventions: Drug: Propofol; Drug: Fentanyl; Drug: Rocuronium bromide

INTERVENTIONS:
Drug: Remimazolam — Lyophilisate for preparation of solution for intravenous administration, 50 mg. Required to prepare a 50 ml syringe with the infusion solution at a concentration of 1 mg/ml (in accordance with guidance given in protocol)
  Arms: Remimazolam
Drug: Propofol — Emulsion for infusion, 10 mg/mL in 20-mL glass vials
  Other Names: Diprivan®
  Arms: Propofol
Drug: Fentanyl — Solution for intravenous administration, 50 mg/mL. Used for anesthesia induction (at a dose of 2 mg/kg) and, if necessary, anesthesia maintenance (the dose was selected individually)
Drug: Rocuronium bromide — Solution for intravenous administration, 10 mg/mL. Used for anesthesia induction (at a dose of 0.6-0.9 mg/kg) and, if necessary, anesthesia maintenance (the dose was selected individually)

SUMMARY:
The purpose of this study was to perform comparative evaluation of clinical efficacy and safety of Remimazolam and Propofol for induction and maintenance of general anesthesia in patients undergoing elective surgery under general anaesthesia.

DETAILED DESCRIPTION:
Only patients with scheduled operations were screened for eligibility in this study. Screening period for each patient lasted from 1 to 14 days. All patients eligible as per protocol criteria were randomized in 1:1 ratio to receive investigational or reference drug. Randomisation was carried out in admission to the operating room - Day1.

For the induction of anesthesia, first there was administration of the trial drug / reference drug, then - administration of a narcotic analgesic (fentanyl at a dose of 2 mg/kg), after which after loss of consciousness, muscle relaxant was used (rocuronium bromide at a dose of 0.6-0.9 mg/kg). Tracheal intubation was performed after achieving the necessary relaxation of the muscles.

Maintenance of anesthesia during surgery was done using the trial drug / reference drug, muscle relaxant (rocuronium bromide - if necessary, during the anesthesia maintenance, the dose was selected individually) and narcotic analgetic (fentanyl, if necessary, during the anesthesia maintenance, the dose was selected individually). To control patient's condition before, during and after surgery, the significant vital parameters were monitored (level of blood pressure and heart rate, respiratory rate, body temperature, saturation, intraoperative ECG, bispectral index (BIS)).

After the operation patients were transferred to the postoperation room where the assessment of the operation memory, and possible presence of postoperative delirium was performed as well as on Day 2. Further treatment and determination of compliance of patient's condition with the criteria for discharge from the hospital was carried out in accordance with current practice of the center.

In 7 (± 2) days after the end of trial drugs administration, patient's condition monitoring and safety evaluation were carried out through telephone contact with the patient, during which data on adverse events and concomitant therapy were collected. Scheduled trial duration for each patient was a maximum of 24 days.

Therapy was considered ineffective, if other sedatives were required for induction (loss of consciousness was not registered after study drugs dose adjustment) and/or maintenance of the required level of sedation during anesthesia (in case of signs of awakening appeared and remained after study drugs dose adjustment).

Therapy efficacy evaluation was based on primary and secondary efficacy criteria. Effect of general anesthetic, a combined evaluation criterion consisted of the following criteria. The trial drug/reference drug was regarded effective in patients who had not had any of the below criteria and ineffective in patients who had at least one of the below criteria:

1. Intraoperative awakening / preservation of memories of operations;
2. The need for additional sedation.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form to participate in the study prior to initiation of any study-related procedures, and possibility to follow the protocol.
2. Body mass index (BMI) calculated as body weight (kg)/height (m)2, ≤ 30 kg/m2.
3. Patients hospitalized for elective surgery in whom intraoperative mechanical ventilation using tracheal intubation (oropharyngeal or nasotracheal) is planned.
4. Patients for whom the duration of inpatient hospital stay for at least 2 days (1 day before and 1 day after the surgery).
5. American Society of Anesthesiologists scale (ASA) I - II functional class.
6. For females: negative result of a pregnancy test (urine test using test strips) since the moment of enrollment to the study prior to administration of the test drug/reference drug, as well as consent to use birth control methods throughout the entire study (since the moment of enrollment to the study until the complete ending of the observation period) for women of childbearing potential.

   Female patients who did not have menstrual periods for 2 years or more before enrollment to the study or female patients who underwent a surgical procedure (surgical sterilization, bilateral oophorectomy, hysterectomy etc.) are considered females of no childbearing potential.
7. For males: consent to use birth control methods throughout the entire study (since the moment of enrollment to the study until the complete ending of the observation period).

Exclusion Criteria:

1. Patients in whom local anesthesia is planned (subarachnoid (spinal) block, epidural anesthesia or peripheral nerve block) during the period from admission into an operating room till extubation on Day 1 (administration of the test drug/reference drug).
2. Patients in whom organ transplantation is planned.
3. Patients in whom heart surgery is planned.
4. Patients with uncontrolled hypertension (e.g. systolic blood pressure ≥160 mm Hg while on antihypertensive therapy).
5. Patients in whom total bilirubin level ≥ 51 mmol/l or aspartate aminotransferase (AST) or alanin aminotransferase (ALT) level ≥ 2.5 upper limit of normal (ULN) (or ≥100 U/L) during the period from Day -14 till their admission to the operating room.
6. Patients in whom serum creatinine level ≥140 mmol/l during the period from Day -14 till their admission to the operating room.
7. Patients undergoing an urgent surgical procedure.
8. Patients in whom a surgical procedure lasting less than 1 hour is planned.
9. Patients in whom extubation problems are anticipated due to the expected necessity of prolonged respiratory support using tracheal intubation.
10. Patients with history of resistance to benzodiazepines or propofol.
11. Patients with history of hypersensitivity to benzodiazepines, propofol, opioid analgesics, fentanyl citrate, rocuronium bromide, sugammadex sodium, flumazenil, naloxone, or other anesthetics or benzodiazepine receptor antagonists.
12. Acute open-angle glaucoma.
13. Myasthenia gravis or myasthenic syndrome.
14. Patients with shock or coma.
15. Acute alcohol intoxication.
16. Patients with epilepsy.
17. Patients with inserted pacemaker with a bioelectric impedance sensor.
18. Patients in whom correct evaluation of the bispectral index (BIS) cannot be performed due to a structural brain disorder.
19. Patients who received benzodiazepines, in case the period between their discontinuation and the administration of the test drug/reference drug is less than 5 half-lives of benzodiazepine (or 5 half-lives of the active metabolites, if applicable), or in case benzodiazepines are revealed in urine test during the screening.
20. Patients taking psychotropic drugs (depot forms should be discontinued at least 1 month prior to the screening; administration of typical forms should be discontinued at least 1 week prior to the screening).
21. Patients in whom massive blood loss is expected (e.g. at least 15% of the circulating volume) during the surgery.
22. History of severe allergic reactions.
23. Alcohol and/or drug abuse or history of such abuse.
24. Nursing women.
25. Patients in whom any other unregistered drugs (including prescription of unregistered combination products or new pharmaceutical forms during the clinical study) are planned within 120 days prior to administration of the study drugs.
26. Patients admitted incapacitated to give an informed consent due to dementia, etc.
27. Patients receiving (had a history of receiving) any medicinal product containing the active substance similar to remimazolam.
28. Patients with exacerbation of existing mental disorders.
29. Patients with a confirmed or suspected malignancy of any localization.
30. Detection of viral hepatitis B and C, HIV infection or syphilis based on the results of screening investigations.
31. Patients considered not conforming to the objectives of this study for any other reasons by the Principal Investigator or the Investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-08-22 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-05-24 (Actual)

PRIMARY OUTCOMES:
ANAESTassessment | During the surgery and 24 hours after the study drugs administration
  "Action as a general anesthetic", a compound evaluation criterion, consisted of the following criteria. The test drug/comparator were considered effective in patients who had not had any of the following criteria and ineffective in patients who had at least one of the following criteria:
  1. Intraoperative awakening/preservation of memories of surgery;
  2. The need for additional sedatives.

SECONDARY OUTCOMES:
TIMEextub | From the moment of discontinuation of the test drug / comparator to restoration of spontaneous breathing and removal of the endotracheal tube on Day 1 of treatment
  Extubation time (minutes)
TIMEopeneyes | From the moment of discontinuation of the test drug / comparator to eye opening on Day 1 of treatment
  Time of eyes opening (minutes). A patient was often asked with a normal voice to open his/her eyes. The time to spontaneous eye opening was recorded.
TIMEunconsc | From the onset of administration of the test drug/comparator to unconsciousness on Day 1 of treatment
  Time of unconsciousness
Bispectral index value (BISx) | Every 5 minutes from admission of a patient to the operating room until transfer from the operating room on Day 1 of treatment
  Bispectral index calculation was carried out automatically by the hardware monitor on electrical activity of the brain and could range from 0 (no electrical activity of the brain) to 100 (clear conscience)
TIMEDOB | From the end of administration of the test drug/comparator to the time when the patient will be able to say the date of his/her birth on Day 1 and 2 of treatment
  Date of birth memory
TIMEORleave | From the end of administration of the test drug/comparator to the time when the patient is transferred from the operating room on Day 1 of treatment
  Operation room leaving time - the time when a patient's condition meets the criteria for transfer from the operating room
TIMErecuper | From the end of administration of the study drug/comparator until the patient reaches the modified Aldrete's system score of ≥9 points on Day 1 of treatment
  Total recovery time assessed by the modified Aldrete scale - a commonly used scale (0-10 points) for determining when patients can be safely discharged from the post-anesthesia care unit assessing patient's activity, respiration, circulation, consciousness and oxygen saturation.

OTHER OUTCOMES:
Number of blood pressure measurement points with systolic blood pressure ≤ 50 mm Hg and ≥ 180 mm Hg | During the surgery
Number of patients needed vasopressor use | During the surgery
  Number of patients developed hypotension during the operation required treatment with vasopressors

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Samsonov, Study Director — R-Pharm
Locations (6):
- Russia (6):
  - FSBI Central Clinical Hospital and Polyclinic of Adminisatration of the President of the Russian Federation, Moscow
  - FSBI Russian National Medical and Surgical Center n.a. N.I.Pirogov, Moscow
  - SBHI City Clinical Hospital №1 n.a. N.I. Pirogov, Moscow
  - SBHI City Clinical Hospital №64 n.a. V.V. Vinogradov, Moscow
  - SBHI Institute of Surgery n.a. A.V.Vishevsky, Moscow
  - SBHI Moscow Clinical Research and Practical center of Department of Healthcare of the city of Moscow, Moscow